CLINICAL TRIAL: NCT04826328
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Efficacy, and Systemic Exposure of a Single Administration of FX301 Via Nerve Block for Management of Post-surgical Pain Following Bunionectomy
Brief Title: Study to Evaluate the Safety and Tolerability of FX301 in Patients Undergoing Bunionectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FX301-2020-001
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative; Bunion
MeSH Terms: conditions — Pain, Postoperative; Bunion | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Part I - Double-Blind, placebo-controlled, three-step, Single Ascending Dose Part II - Double Blind, placebo-controlled, Expansion Phase to enroll additional patients to an SMC-cleared dose/volume level
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- FX301 Low Dose Low Volume (Experimental): 65 mg of funapide given as a single injection nerve block adjacent to the sciatic nerve of the popliteal fossa
  Interventions: Drug: FX301
- FX301 Low Dose High Volume (Experimental): 130 mg of funapide given as a single injection nerve block adjacent to the sciatic nerve of the popliteal fossa
  Interventions: Drug: FX301
- FX301 High Dose Low Volume (Experimental): 130 mg of funapide given as a single injection nerve block adjacent to the sciatic nerve of the popliteal fossa
  Interventions: Drug: FX301
- FX301 High Dose High Volume (Experimental): 260 mg of funapide given as a single injection nerve block adjacent to the sciatic nerve of the popliteal fossa
  Interventions: Drug: FX301
- Normal Saline (Placebo Comparator): Low or high matching volume of preservative-free normal saline given as a single injection adjacent to the sciatic nerve of the popliteal fossa
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: FX301 — FX301 is an extended-release formulation of funapide being developed as a single injection peripheral nerve block for the management of acute postsurgical pain
  Other Names: funapide
  Arms: FX301 High Dose High Volume; FX301 High Dose Low Volume; FX301 Low Dose High Volume; FX301 Low Dose Low Volume
Drug: Normal Saline — Single peripheral nerve injection
  Arms: Normal Saline

SUMMARY:
This two-part study will be conducted in male and female patients 18 to 65 years of age undergoing bunionectomy.

Part I - three-step, single ascending dose study design in which two drug loads (low drug load of funapide and high drug load of funapide) and two volumes (high volume and low volume) of FX301 will be explored against placebo in four cohorts of 12 patients each (9 active:3 placebo) for the management of post-surgical pain in patients undergoing bunionectomy.

Part II - expansion cohort to further assess safety, tolerability, systemic exposure, and efficacy of a selected drug load/volume of FX301. An additional 36 patients will be randomized in a 1:1 ratio to receive either FX301 or placebo as a single-injection analgesic nerve block adjacent to the sciatic nerve of the popliteal fossa.

DETAILED DESCRIPTION:
This two-part study will be conducted in male and female patients 18 to 65 years of age undergoing bunionectomy.

Part I - three-step, single ascending dose study design in which two drug loads (low drug load of funapide and high drug load of funapide) and two volumes (high volume and low volume) of FX301 will be explored against placebo in four cohorts of 12 patients each (9 active:3 placebo) for the management of post-surgical pain in patients undergoing bunionectomy. At each step, the amount of FX301 administered (dose level) will be constant (65 mg, 130 mg, and 260 mg) so that the local safety of the drug loads and the volumes administered can be assessed separately. The 130 mg dose step will consist of both the low drug load at high volume and the high drug load at low volume concentrations.

A Safety Monitoring Committee (SMC) will review all safety data of each dose step prior to escalation to the next dose level.

After completion of the last cohort, data will be reviewed to assess whether to expand one of the four dose/volume cohorts up to and including the highest tolerated drug load/volume.

Part II - expansion cohort to further assess safety, tolerability, systemic exposure, and efficacy of a selected drug load/volume of FX301. An additional 36 patients will be randomized in a 1:1 ratio to receive either FX301 or placebo as a single-injection analgesic nerve block adjacent to the sciatic nerve of the popliteal fossa.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate in the study
2. Be willing and able to complete study procedures and pain scales, follow instructions and communicate meaningfully in English with study personnel, and return for outpatient follow-up visits as required.
3. Male or female ≥18 to ≤65 years of age, inclusive
4. Planning to undergo an elective primary unilateral, distal, first metatarsal bunionectomy with osteotomy and internal fixation, without collateral procedure or additional surgeries, to be performed under Monitored Anesthesia Care (MAC) and be eligible to receive a popliteal sciatic nerve block
5. Classified as either ASA 1 or ASA 2 by the American Society of Anesthesiologists Physical Status Classification System (Appendix 1).
6. Has a BMI of ≥18 to ≤ 35 kg/m2.
7. Willing to washout from all prohibited medications for the longer of 14 days or five half-lives prior to dosing, and abstain from those medications through the end of study (Appendix 5).
8. If a male, unless he has a same sex partner, be either sterile (surgically or biologically) or commit to an acceptable method of birth control while participating in the study.
9. If a woman of childbearing potential (WOCBP), must meet all of the following:

   * Not be pregnant (WOCBP must have a negative serum pregnancy test at screening and negative urine pregnancy test before surgery);
   * Not plan to become pregnant or to breast feed during the study; and
   * Be surgically sterile (at least one year post total hysterectomy, bilateral oophorectomy or bilateral tubal ligation) or at least one year post-menopausal, have a monogamous partner who is surgically sterile, have a same sex partner, or (one of the following must apply):

     * is practicing double-barrier contraception
     * is practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity)
     * is using a non-hormonal contraceptive approved by the FDA for at least 2 months prior to screening and commits to the use of an acceptable form of birth control while participating in the study..

Exclusion Criteria:

1. Has a concurrent painful condition, other than bunion-related pain, that may require analgesic treatment during the study period or may confound post-surgical pain assessments.
2. Has an active skin disease or other clinically significant abnormality at the anticipated site of surgery or nerve block insertion site that could interfere with the planned surgery.
3. Has had previous bunionectomy or other surgical procedure on the index foot that could impact the current bunion surgery.
4. Has any clinically significant cardiac, respiratory, neurological, immunological, hematological, or renal disease or any other condition that, in the opinion of the investigator, could compromise the subject's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
5. Has a known history of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, opioids, or any NSAIDs; history of NSAID-induced bronchospasm (subjects with the triad of asthma, nasal polyps, and chronic rhinitis are at greater risk for bronchospasm and should be considered carefully); or hypersensitivity, allergy, or significant reaction to any other drugs used in the study, including anesthetics and antibiotics that may be required on the day of surgery.
6. Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
7. Has taken any opioids, NSAIDS, or acetaminophen within 3 days prior to the scheduled surgery. Low dose aspirin (<100 mg) for cardiovascular protection is acceptable.
8. Has initiated treatment with any of the following medications within 30 days prior to study medication administration or is taking any of these medications to control pain: selective serotonin reuptake inhibitors, selective norepinephrine reuptake inhibitors, gabapentin, pregabalin, or cyclooxygenase-2 inhibitors. (Note: If a subject is taking one of these medications for a reason other than pain control, the subject must be on a stable scheduled dose [i.e., not "as needed"] for at least 1 month prior to study medication administration.)
9. Within the 14 days prior to surgery, be taking parenteral or oral corticosteroids (steroid inhalers for allergy or asthma treatment, topical steroids for a non-clinically significant skin condition not involving the area of surgery, or ophthalmic steroids are permissible).
10. Is currently receiving antianginal therapy
11. Has a known or suspected history of alcoholism or drug abuse or misuse within 1 year of screening or evidence of opioid tolerance or physical dependence before dosing with the study medication.
12. Has positive results on the alcohol test (breath or saliva) indicative of alcohol abuse or urine drug screen (UDS) indicative of illicit drug use at screening, and/or prior to surgery. Note that for those subjects have a history of, or who test positive for tetrahydrocannabinol (THC), if they are willing to abstain from use or consumption of THC-containing products from 14 days prior to surgery to Day 85, they may be allowed to participate in the study. Additionally, it may be permissible for the subject to participate if the results of the UDS can be explained by a current prescription or acceptable over-the-counter medication as determined by the investigator at screening and/or prior to surgery.
13. Has significant difficulties swallowing tablets or is unable to tolerate oral medication.
14. Has received any investigational drug or device or investigational therapy within the last 30 days.
15. Has a history of a clinically significant (in the investigator's opinion) GI event within 6 months before screening or has any history of peptic or gastric ulcers or GI bleeding.
16. Has a surgical or medical condition of the GI or renal system that might significantly alter the absorption, distribution, or excretion of any drug substance.
17. Is considered by the investigator to be an unsuitable candidate to receive the study medication for any reason (including, but not limited to, the risks described as precautions, warnings, and contraindications in the current version of the IB).
18. Is receiving systemic chemotherapy, has an active malignancy of any type, or has been diagnosed with cancer within 2 years before screening (excluding squamous or basal cell carcinoma of the skin that has been clinically stable and/or fully excised in a curative procedure).
19. Has significant renal disease, as indicated by clinical laboratory assessment (creatinine > 1.9 mg/dL).
20. Has significant hepatic disease, as indicated by clinical laboratory assessment (results ≥ 2 times the upper limit of normal for any liver function test (LFT), including aspartate aminotransferase (AST), alanine aminotransferase (ALT), and lactate dehydrogenase (LDH)).
21. Has a known history of seizure disorder, a family history of seizures, or previous head trauma.
22. Has loss of sensation in extremities or significant peripheral neuropathy.
23. Laboratory evidence of infection with HIV, positive test for HBsAg, or positive serology for hepatitis C virus (HCV) with positive test for HCV RNA.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events after FX301 is administered as a single-dose, analgesic nerve block | Baseline to Day 85
  Incidence of treatment emergent adverse events after a single analgesic nerve block of FX301

SECONDARY OUTCOMES:
Efficacy of FX301 in the management of acute post-surgical pain | Baseline to 72 Hours
  Sum of pain intensity as measured by Numeric Rating Scale (NRS) from 0 to 10, 0 being no pain and 10 being the worst pain imaginable
Characterization of the systemic exposure of funapide as seen through the pharmacokinetic (PK) analysis at Days 1-6, 8, 15, 29, 57, and 85. | Baseline to Day 85
  Measure of the concentration of funapide in blood plasma and urine

CONTACTS AND LOCATIONS:
Overall Officials: William T Andrews, MD, FACP, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- Lotus Clinical Research, Huntington Hospital, Pasadena, California, United States